CLINICAL TRIAL: NCT03885167
Title: Identification of Biomarkers in Spinocerebellar Ataxia 3
Acronym: SCA3
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Henry Paulson, Professor of Neurology, University of Michigan
Other Study IDs: HUM00121991; U01NS106670 (NIH)
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Spinocerebellar Ataxia Type 3
MeSH Terms: conditions — Machado-Joseph Disease | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Approximately 2 tablespoons (approximately 30 ml) of CSF will be collected, along with a single collection of about 3.5 tablespoons (approximately 50 ml) of blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected Individuals with Known SCA3: In order to be eligible for this cohort, participants must have confirmed genetic testing results for Spinocerebellar Ataxia Type 3.
  Interventions: Other: Specimen Collection
- Healthy Individual Control Subjects: In order to be eligible for this cohort, subjects must not have a diagnosis of Spinocerebellar Ataxia Type 3 and no major medical issues including but not limited to conditions that would cause an unsafe specimen collection.
  Interventions: Other: Specimen Collection

INTERVENTIONS:
Other: Specimen Collection — No interventions take place as part of study participation- only specimen collection occurs for both cohorts.

SUMMARY:
The purpose of this study is to examine the differences in cerebral spinal fluid (CSF) and blood of patients with spinocerebellar ataxias and healthy volunteers. The goal of this project is to identify new biomarkers that are useful for characterizing spinocerebellar ataxias and identify targets for treatment or prevention of this condition.

DETAILED DESCRIPTION:
Participants will undergo a SARA exam, a lumbar puncture and a blood draw. A lumbar puncture is a procedure in which a small amount of the spinal fluid that surrounds the brain and spinal cord is removed by inserting a needle in the lower back. Participants will be asked not to eat or drink anything (water is acceptable) for at least 6 hours before the lumbar puncture visit. For this procedure, participants will be positioned lying on their side and curled up in a ball, or sitting up and bent forward, whichever is easier. Cushions will be used to enhance comfort. The lower back region will be cleaned and disinfected with an antiseptic iodine solution. The doctor will inject local anesthetic (lidocaine, 1%) into the skin of the lower back. This may produce a transient, mild burning sensation. A very small needle will be introduced into the skin and moved into fluid-filled space around the spinal nerves coming from the spinal cord. This may produce a pressure sensation. Approximately 2 tablespoons approximately 30 ml) of fluid will be collected. The needle will be removed and a band-aid applied over the needle insertion site. Participants will be asked to remain stationary, lying on flat for about ½ hour on a bed in the research clinic. Participants will be given something to eat and drink before leaving. Strenuous physical activity should be avoided for the next 24 hours. This includes lifting, bending, doing housework and gardening, or doing exercise such as jogging or bicycle riding. The SARA (Scale for the Assessment and Rating of Ataxia) exam is a clinical scale that assesses a range of different impairments in cerebellar ataxia. The scale is made up of 8 items related to gait, stance, sitting, speech, fingerchase test, nose-finger test, fast alternating movements and heel-shin test, and takes approximately 15 minutes to complete.

The study also involves a single collection of about 3.5 tablespoons (approximately 50 ml) of blood. This blood draw may take place during a regularly scheduled visit to the neurology clinic or at the research appointment.

ELIGIBILITY:
Inclusion Criteria:

•Confirmed Genetic Testing of SCA3 or Healthy Volunteers

Exclusion Criteria:

* People with:

  * unstable thyroid
  * unstable intestinal/stomach issues
  * unstable heart issues
  * unstable liver issues
  * unstable kidney issues
  * unstable lung issues
  * unstable hormone issues
  * unstable mental disorders at screening
  * a tumor or evidence of having a tumor
  * a chronic infection or any severe acute infection within 3 months prior to screening
* People who:

  * Take anti-coagulants and NSAIDs
  * Have started any investigational medications in the last month
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Within the local community and/or those associated with the National Ataxia Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Change in Ataxin 3 Levels in Cerebrospinal Fluid Specimens | 4 Hours
  A lumbar puncture is performed to collect CSF.
Change in Ataxin 3 Levels in Blood Plasma Specimens | 4 Hours
  A single blood draw is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Paulson, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
At this time, no specific description of a sharing plan was incorporated into the approved grant, and there are no requirements that pertain to this action. Therefore, until more information is obtained as the study progresses, there is no plan to share at this time.